CLINICAL TRIAL: NCT00615550
Title: The Effect of Vaginal Progesterone Administration in the Prevention of Preterm Birth in Women With a Short Cervix [Vaginal Progesterone Bioadhesive Gel (Prochieve)® Extending Gestation A New Therapy for Short Cervix - Trial (PREGNANT Short Cervix - Trial)]
Brief Title: PREGNANT Short Cervix Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Juniper Pharmaceuticals, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COL-1620-302; 09-CH-N014
Record Dates: First submitted 2008-01-18; First posted 2008-02-14 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-02

CONDITIONS: Preterm Delivery; Short Cervix; Short Uterine Cervical Length
Keywords: Preterm; Cervix
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo vaginal gel
  Interventions: Drug: placebo
- Prochieve (Active Comparator): Progesterone 8% Vaginal Gel
  Interventions: Drug: progesterone

INTERVENTIONS:
Drug: progesterone — 8% vaginal gel, 1.125 Grams once daily, beginning at 19 0/7 to 23 6/7 weeks gestation through 36 6/7 weeks gestation
  Other Names: Prochieve 8%
  Arms: Prochieve
Drug: placebo — vaginal gel, 1.125 Grams once daily, beginning at 19 0/7 to 23 6/7 weeks gestation through 36 6/7 weeks gestation
  Arms: Placebo

SUMMARY:
The purpose of this research study is to evaluate the usefulness of progesterone vaginal gel in decreasing the preterm birth rate in a population of pregnant women with short cervical length and at high risk for preterm birth.

DETAILED DESCRIPTION:
A Short uterine cervical length in the mid-trimester is the most powerful predictor of preterm birth.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a short cervical length by transvaginal ultrasound (TVU) defined as 10-20mm. In cases of "dynamic cervix", the shortest observed/documented cervical length by TVU is to be used as the cervical length for inclusion purposes.
2. Singleton gestation.
3. The pregnancy has an estimated gestational age between 19 0/7 weeks and 23 6/7 weeks.
4. Maternal age between 15 (or local age of majority/emancipation) and 45 years of age at the time of screening. An alternative age range can be accepted according to the standards and applicable regulations of the study centers.
5. The subject speaks either English or a common local language.
6. The subject has voluntarily signed the Informed Consent Form and associated forms after having the contents explained, and all her questions are answered to her satisfaction and understanding.
7. In the opinion of the investigator, the subject is able to understand the study and is able to give informed consent, as well as participate in it and adhere to study procedures.

Exclusion Criteria:

1. The subject has a cervical length <10 or >20mm.
2. The subject has a multifetal gestation.
3. The subject has or is scheduled to have a cervical cerclage prior to randomization. According to ACOG Practice Bulletin Number 48 (November 2003), cerclage can be considered in a subject with a history of 3 or more unexplained midtrimester pregnancy losses or preterm deliveries.228,229
4. Subjects diagnosed to have acute cervical insufficiency with bulging membranes passing the external os.
5. The subject has a previous history of an adverse reaction to progesterone or any component present in Prochieve® 8% vaginal gel.
6. The subject has been treated with a progestogen within the previous 4 weeks.
7. The subject is currently being treated for a seizure disorder, has an unstable psychiatric disorder, is taking antihypertensive therapy for chronic hypertension at the time of enrollment, has a history of congestive heart failure or chronic renal failure, or has uncontrolled diabetes mellitus (known end-organ dysfunction secondary to vascular disease).
8. The subject has active thrombophlebitis or a thromboembolic disorder, or a history of hormone-associated thrombophlebitis or thromboembolic disorders.
9. The subject has active liver dysfunction or disease.
10. The subject has known or suspected malignancy of the breast or genital organs.
11. The subject is currently participating in another interventional study or has participated in an interventional drug study within one month prior to screening for this study.
12. The subject's current pregnancy is complicated by a major fetal anomaly or known chromosomal abnormality.
13. The subject has a uterine anatomic malformation (bicornuate uterus, septate uterus)
14. The subject, in the judgment of the investigator, will be unable or unwilling to comply with study-related assessments and procedures.
15. The subject currently has preterm rupture of membranes, vaginal bleeding, known or suspected amnionitis, or signs or symptoms of preterm labor at the time of enrollment.
16. The subject is HIV positive with a CD4 count of <350 cells/mm3 and is receiving more than one (1) medication to prevent the transfer of AIDS to the fetus.
17. Complete placenta previa.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 465 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George W. Creasy, MD, FACOG, Study Director — Columbia Laboratories, Inc.; Roberto Romero, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Sonia Hassan, MD, Study Director — Wayne State University
Locations (49):
- United States (27):
  - University of South Alabama Dept. of OB/GYN, Mobile, Alabama
  - St. Joseph's Hospital and Med Ctr Women's Care Center, Phoenix, Arizona
  - UCI Medical Center, Orange, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Miami Leonard Miller School of Medicine Department of Obstetrics and Gynecology, Miami, Florida
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Perinatal Center of Iowa, Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Perinatal Diagnostic Center, Lexington, Kentucky
  - Johns Hopkins Community Physicians, Baltimore, Maryland
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Perinatology Research Branch Hutzel Women's Hospital, Detroit, Michigan
  - Henry Ford Healthcare System, Detroit, Michigan
  - Spectrum Health Research Department, Grand Rapids, Michigan
  - St. Joseph Mercy-Oakland, Pontiac, Michigan
  - Washington University School of Medicine, Dept. of OB/GYN, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Winthrop University Hosital, Mineola, New York
  - Albert Einstein Hospital, The Bronx, New York
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - UPHS Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital OB/GYN / Maternal Fetal Medicine, Philadelphia, Pennsylvania
  - Regional Obstetrical Consultants, Chattanooga, Chattanooga, Tennessee
  - Regional Obstetrical Consultants, Knoxville, Knoxville, Tennessee
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Charleston Area Medical Center Clinical Trials Center, Charleston, West Virginia
- Belarus (2):
  - 1st Clinical Hospital of the City of Minsk, Minsk
  - Public Health Services Establishment "Vitebsk City Clinical Hospital of First Aid", Vitebsk
- Chile (2):
  - Escuela De Medicina, Pontificia Universidad Catolica De Chile, Santiago
  - Maternidad Hospital DR Sotero Del Rio, Santiago
- Charles University & General Teaching Hospital, Prague, Czechia
- India (5):
  - BJ Medical College & Sassoon Hospital, Pune, Maharashtra
  - Sri Ramchandra Medical College and Research Institute, Porur, Tamil Nadu
  - Sheth L.G. Hospital, Ahmedabad
  - MediCiti Institute of Medical Sciences, Andhra Pradesh
  - Government Medical College, Nagpur
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Kaplan Medical Center, Rehovot
  - Sheba Medical Center, Tel Litwinsky
- Azienda Ospedaliera di Padova Centro Prenatale Divisione di Ostetricia, Padua, Italy
- Russia (2):
  - Limited Liability Company "American Health Clinic", Saint Petersburg
  - Saint Petersburg State Healthcare Institution Maternity Hospital 17, Saint Petersburg
- Steve Biko Academic Hospital Dept. of OB-GYN and Maternal Fetal Medicine, Pretoria, South Africa
- Ukraine (5):
  - Municipal health care establishment "City Maternity Clinical Hospital", Chernivtsi
  - Department of Obstetrics and Gynecology of Dnepropetrovsk State Medical Academy, Municipal establishment "City Maternity Hospital # 1", Dnipro
  - M. Gorky Donetsk National Medical University, Department of Obstetrics, Gynecology and Perinatology, Maternity Hospital of 6th Central City Clinical Hospital, Donetsk
  - Municipal clinical hospital #1, Kiev
  - Antenatal Clinic # 1, Central Polyclinics of Pechersk District, Kyiv

REFERENCES:
- [Background] O'Brien JM, Adair CD, Lewis DF, Hall DR, Defranco EA, Fusey S, Soma-Pillay P, Porter K, How H, Schackis R, Eller D, Trivedi Y, Vanburen G, Khandelwal M, Trofatter K, Vidyadhari D, Vijayaraghavan J, Weeks J, Dattel B, Newton E, Chazotte C, Valenzuela G, Calda P, Bsharat M, Creasy GW. Progesterone vaginal gel for the reduction of recurrent preterm birth: primary results from a randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2007 Oct;30(5):687-96. doi: 10.1002/uog.5158. PMID 17899572
- [Background] DeFranco EA, O'Brien JM, Adair CD, Lewis DF, Hall DR, Fusey S, Soma-Pillay P, Porter K, How H, Schakis R, Eller D, Trivedi Y, Vanburen G, Khandelwal M, Trofatter K, Vidyadhari D, Vijayaraghavan J, Weeks J, Dattel B, Newton E, Chazotte C, Valenzuela G, Calda P, Bsharat M, Creasy GW. Vaginal progesterone is associated with a decrease in risk for early preterm birth and improved neonatal outcome in women with a short cervix: a secondary analysis from a randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2007 Oct;30(5):697-705. doi: 10.1002/uog.5159. PMID 17899571
- [Background] Fonseca EB, Celik E, Parra M, Singh M, Nicolaides KH; Fetal Medicine Foundation Second Trimester Screening Group. Progesterone and the risk of preterm birth among women with a short cervix. N Engl J Med. 2007 Aug 2;357(5):462-9. doi: 10.1056/NEJMoa067815. PMID 17671254
- [Background] Romero R. Prevention of spontaneous preterm birth: the role of sonographic cervical length in identifying patients who may benefit from progesterone treatment. Ultrasound Obstet Gynecol. 2007 Oct;30(5):675-86. doi: 10.1002/uog.5174. No abstract available. PMID 17899585
- [Result] Hassan SS, Romero R, Vidyadhari D, Fusey S, Baxter JK, Khandelwal M, Vijayaraghavan J, Trivedi Y, Soma-Pillay P, Sambarey P, Dayal A, Potapov V, O'Brien J, Astakhov V, Yuzko O, Kinzler W, Dattel B, Sehdev H, Mazheika L, Manchulenko D, Gervasi MT, Sullivan L, Conde-Agudelo A, Phillips JA, Creasy GW; PREGNANT Trial. Vaginal progesterone reduces the rate of preterm birth in women with a sonographic short cervix: a multicenter, randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2011 Jul;38(1):18-31. doi: 10.1002/uog.9017. Epub 2011 Jun 15. PMID 21472815
- [Result] Romero R, Nicolaides K, Conde-Agudelo A, Tabor A, O'Brien JM, Cetingoz E, Da Fonseca E, Creasy GW, Klein K, Rode L, Soma-Pillay P, Fusey S, Cam C, Alfirevic Z, Hassan SS. Vaginal progesterone in women with an asymptomatic sonographic short cervix in the midtrimester decreases preterm delivery and neonatal morbidity: a systematic review and metaanalysis of individual patient data. Am J Obstet Gynecol. 2012 Feb;206(2):124.e1-19. doi: 10.1016/j.ajog.2011.12.003. Epub 2011 Dec 11. PMID 22284156
- See also: Ultrasound Obstet Gynecol (2011) — http://onlinelibrary.wiley.com/doi/10.1002/uog.9017/pdf
- See also: Open Access to Final Study Result Publication — http://onlinelibrary.wiley.com/doi/10.1002/uog.9017/pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2008 to June 2010
Period: Overall Study
Arm/Group | Placebo | Prochieve
Started | 229 | 236
Completed | 223 | 235
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Prochieve | Total
Number analyzed (Participants) | 223 | 235 | 458
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 223 | 235 | 458
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.1) | 26.5 (5.8) | 26.4 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 235 | 458
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belarus | 7 | 5 | 12
  United States | 100 | 107 | 207
  Czech Republic | 1 | 3 | 4
  Ukraine | 26 | 28 | 54
  South Africa | 11 | 10 | 21
  Russian Federation | 0 | 1 | 1
  Israel | 0 | 3 | 3
  Chile | 2 | 0 | 2
  Italy | 3 | 5 | 8
  India | 73 | 73 | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Birth <=32 6/7 Weeks Gestation.
Time Frame: 9 to 13 weeks
Population: Intent to Treat
Measure: Number; unit: participants
Arm/Group | Placebo | Prochieve
Number analyzed (Participants) | 223 | 235
participants | 36 | 21
Statistical Analysis 1: Comparison: Placebo vs Prochieve; Test type: Superiority or Other; p = 0.020, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.55, 95% CI 2-sided [0.33 to 0.92]

2. Secondary Outcome: Number of Infants With Neonatal Morbidities Such as Respiratory Distress Syndrome (RDS), Bronchopulmonary Dysplasia (BPD), Intraventricular Hemorrhage (IVH), Proven Sepsis, and Necrotizing Enterocolitis (NEC)
Description: Each infant is scored based on the 7 morbidity and mortality events above:
  0= no morbidity event
  1. 1 morbidity event
  2. 2 morbidity events
  3. 3 or more morbidity events
  4. mortality
Time Frame: Delivery Hospitalization (1-212 days)
Measure: Number; unit: participants
Arm/Group | Placebo | Prochieve
Number analyzed (Participants) | 223 | 235
participants
  Composite score 0 | 192 | 217
  Composite score 1 | 11 | 5
  Composite score 2 | 8 | 2
  Composite score 3 | 0 | 3
  Composite score 4 | 11 | 8
  Infants with RDS | 17 | 7
Statistical Analysis 1: Comparison: Placebo vs Prochieve; Statistical analysis presented for composite score data; Test type: Superiority or Other; p = 0.048, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Prochieve; Statistical analysis presented for RDS data; Test type: Superiority or Other; p = 0.026, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.39, 95% CI 2-sided [0.17 to 0.92]

3. Secondary Outcome: Number of Subjects With Preterm Birth at ≤27 6/7, ≤34 6/7, and <36 6/7 Weeks Gestation.
Description: Number of participants at <=27 6/7 , <=34 6/7, and <36 6/7.
Time Frame: Gestational Age at Delivery
Population: Intent to Treat
Measure: Number; unit: participants
Arm/Group | Placebo | Prochieve
Number analyzed (Participants) | 223 | 235
participants
  Number of deliveries <= 27 6/7 weeks | 23 | 12
  Number of deliveries <= 34 6/7 weeks | 52 | 34
  Number of deliveries <= 36 weeks | 76 | 71
Statistical Analysis 1: Comparison: Placebo vs Prochieve; Statistical analysis presented for births <=27 6/7 weeks data; Test type: Superiority or Other; p = 0.036, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.5, 95% CI 2-sided [0.25 to 0.97]
Statistical Analysis 2: Comparison: Placebo vs Prochieve; Statistical analysis presented for <= 34 6/7 weeks data; Test type: Superiority or Other; p = 0.016, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.62, 95% CI 2-sided [0.42 to 0.92]
Statistical Analysis 3: Comparison: Placebo vs Prochieve; Statistical analysis presented for <36 weeks data; Test type: Superiority or Other; p = 0.376, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.68 to 1.16]

4. Secondary Outcome: Number of Neonates Who Died.
Time Frame: Delivery to 28 days
Population: All infants with a known delivery date and status.
Measure: Number; unit: participants
Arm/Group | Placebo | Prochieve
Number analyzed (Participants) | 223 | 235
participants | 5 | 3
Statistical Analysis 1: Comparison: Placebo vs Prochieve; Test type: Superiority or Other; p = 0.431, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.57, 95% CI 2-sided [0.14 to 2.35]

5. Secondary Outcome: Number of Infants With a Birth Weight < 1500 Grams or < 2500 Grams
Description: Assessment of birth weight < 1500 grams or < 2500 grams
Time Frame: date of delivery
Population: Available birth weight.
Measure: Number; unit: participants
Arm/Group | Placebo | Prochieve
Number analyzed (Participants) | 220 | 234
participants
  Birth weight < 1500 grams | 30 | 15
  Birth weight < 2500 grams | 68 | 60
Statistical Analysis 1: Comparison: Placebo vs Prochieve; Statistical analysis for birth weight < 1500 grams data; Test type: Superiority or Other; p = 0.01, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.47, 95% CI 2-sided [0.26 to 0.85]
Statistical Analysis 2: Comparison: Placebo vs Prochieve; Statistical analysis for birth weight < 2500 grams data; Test type: Superiority or Other; p = 0.213, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.62 to 1.11]

ADVERSE EVENTS:
Time Frame: Randomization to delivery (1 day to 168 days)
Arm/Group | Placebo | Prochieve
Serious Adverse Events (participants affected / at risk) | 98/224 | 97/235
Other Adverse Events (participants affected / at risk) | 24/223 | 30/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=224) | Prochieve (N=235)
premature baby (Pregnancy, puerperium and perinatal conditions) | 46 (46) | 44 (44)
premature labor (Pregnancy, puerperium and perinatal conditions) | 33 (33) | 17 (17)
premature rupture of the membranes (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 12 (12)
cervix disorder (Reproductive system and breast disorders) | 12 (12) | 21 (21)
uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 5 (5)
foetal distress abnormal (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 6 (6)
cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4)
pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 2 (2)
stillbirth (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3)
chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2)
foetal growth retardation (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1)
pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4)
premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1)
foetal heart rate deceleration (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
funisitis (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
bradycardia foetal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
breech presentation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
cholestasis of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
foetal movements decreased (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
obstructed labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
placenta accreta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
tachycardia foetal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
uterine pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
cervix cerclage procedure (Surgical and medical procedures) | 5 (5) | 9 (9)
maternal therapy to enhance foetal lung maturity (Surgical and medical procedures) | 1 (1) | 1 (1)
abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
ureaplasma infection (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
pyrexia (General disorders) | 2 (2) | 0 (0)
cholecysitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
feotal monitoring (Investigations) | 0 (0) | 1 (1)
gestational diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
physical assault (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=223) | Prochieve (N=235)
abdominal pain (Gastrointestinal disorders) | 11 (11) | 13 (13)
Dyspepsia (Gastrointestinal disorders) | 12 (12) | 15 (15)
Nausea (Gastrointestinal disorders) | 23 (23) | 23 (23)
Vaginitis bacterial (Infections and infestations) | 6 (6) | 12 (12)
Vulvovaginal mycotic infection (Infections and infestations) | 11 (11) | 17 (17)
Headache (Nervous system disorders) | 18 (18) | 16 (16)
Bleeding peripartum (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 9 (9)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 10 (10)
Vaginal infection (Reproductive system and breast disorders) | 11 (11) | 15 (15)
cervix disorder (Reproductive system and breast disorders) | 17 (17) | 23 (23)
anaemia (Blood and lymphatic system disorders) | 14 (14) | 15 (15)
chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 12 (12)
back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 12 (12)
gestational diabetes (Metabolism and nutrition disorders) | 9 (9) | 14 (14)
premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 13 (13)
urinary tract infection (Infections and infestations) | 9 (9) | 11 (11)
foetal growth retardation (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 5 (5)

LIMITATIONS AND CAVEATS:
Trial not powered for subgroup analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No